CLINICAL TRIAL: NCT07335120
Title: A reaL-world Data and Sample coMpendium of frAil aNd/or Multiply treAted Patients With Large B-Cell Lymphoma
Brief Title: A Real-world Data and Sample Compendium of Frail and/or Multiply Treated Large B-cell Lymphoma
Acronym: ALMANAC
Status: Recruiting | Type: Observational
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C1469A; 337564 (Other: IRAS)
Record Dates: First submitted 2026-01-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: DLBCL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, PBMCs, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients with LBCL requiring treatment but considered unsuitable for standard of care (SOC) treatments (full dose R-CHOP or Pola-R-CHP).
- Cohort B: Patients with relapsed/refractory LBCL.

SUMMARY:
LBCL is a cancer of the lymphatic system where B-cells (a type of white blood cell) experience uncontrolled growth. The standard treatment for LBCL is a combination of chemotherapy and immunotherapy, referred to as chemo-immunotherapy. Currently, the best results in the treatment of LBCL is with a chemo-immunotherapy combination called R-CHOP or Pola-R-CHP. Full doses of treatment are not suitable for elderly or frail patients due to potential to cause side effects and heart problems. Such patients either receive a reduced dose called mini-R-CHOP or receive alternatives (e.g. R-GCVP or R-CEOP). Additionally, some patients treated with R-CHOP or Pola-R-CHP may not respond or may respond initially before relapsing. For these patients, treatment is not standardised, and practice varies between hospitals. ALMANAC aims to collect data about the management and outcomes of patients with LBCL who are unsuitable for standard treatments because they are not well enough to tolerate the side effects or because they have not responded or relapsed following initial treatment. In doing so, it will guide research into LBCL leading to a better understanding of this condition and better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects ≥16 years of age at the time of enrolment.
* Ability to understand and sign written informed consent.
* Previously untreated histologically proven Large B-cell non-Hodgkin's lymphoma (LBCL) according to the current World Health Organisation 2016 classification including all morphological variants.

Cohort A:

* Large B-cell lymphomas i) Diffuse large B-cell lymphoma, NOS ii) T-cell/histiocyte-rich large B-cell lymphoma iii) Diffuse large B-cell lymphoma/ high grade B-cell lymphoma with MYC and BCL2 re-arrangements. iv) High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements v) ALK-positive large B-cell lymphoma vi) Large B-cell lymphoma with IRF4 rearrangement vii) High-grade B-cell lymphoma with 11q aberrations or Burkitt-like lymphoma with 11q aberration viii) EBV-positive diffuse large B-cell lymphoma EBV-positive diffuse large B-cell lymphoma, NOS ix) Diffuse large B-cell lymphoma associated with chronic inflammation x) Fibrin-associated large B-cell lymphoma xi) Plasmablastic lymphoma xii) Primary large B-cell lymphoma of immune-privileged sites (vitro-retinal and testis but not CNS) and Intravascular large B-cell lymphoma xiii) Primary mediastinal large B-cell lymphoma xiv) Mediastinal grey zone lymphoma B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classic Hodgkin lymphoma xv) High-grade B-cell lymphoma, NOS xvi) HIV or KSHV/HHV8-positive diffuse large B-cell lymphoma
* De novo presentations of transformed indolent B-cell lymphomas.
* LBCL patients with de novo disease unfit for full dose R-CHOP/Pola-R-CHP OR

Cohort B:

* LBCL patients (as in Cohort A) with relapsed/refractory disease (including de novo transformed indolent B-cell lymphomas) following frontline (one previous line of chemo-immunotherapy) including any line CAR-T therapy.
* Patients fulfilling the above criteria who are on other trials/studies are eligible for recruitment.
* Patients previously registered into Cohort A with subsequent relapsed/refractory disease. Such patients can be registered into cohort B and will be given a new study number that is linked to their study number for cohort A.
* Data for patients commencing treatment <6 months prior to enrolment and with ongoing follow-up can be entered retrospectively.

Exclusion Criteria:

1. Patients treated >6 months prior to trial enrolment (Cohort B).
2. Patients eligible for full dose R-CHOP/Pola-R-CHP (Cohort A)
3. Patients with CNS lymphoma
4. Lymphoid proliferations and lymphomas associated with immune suppression and dysregulation. (e.g., Post-Transplant Lymphoproliferative Disorders)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and female subjects ≥16 years of age at the time of enrolment. Ability to understand and sign written informed consent. Previously untreated histologically proven Large B-cell non-Hodgkin's lymphoma (LBCL) according to the current World Health Organisation 2016 classification including all morphological variants.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints (Cohorts A and B)- Progression Free Survival at 12 months (PFS12): | 12 Month
  Progression Free Survival at 12 months (PFS12): Progression-free survival defined as disease progression or recurrence, or death from any cause, (defined as days from the date of cohort assignment to event) occurring within 12 months as assessed by the investigator using the revised Lugano response criteria for malignant lymphoma (2016).

CONTACTS AND LOCATIONS:
Locations (1):
- The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom